CLINICAL TRIAL: NCT02896049
Title: Celsius TCS Hyperthermia System Post Market Clinical Follow-Up (PMCF) Trial - Vigilance Registry
Brief Title: Celsius TCS Hyperthermia System PMCF Trial
Status: Withdrawn | Type: Observational
Why Stopped: no inclusion has been performed
Sponsor: Celsius42 GmbH (Industry)
Collaborators: Aix Scientifics (Industry)
Responsible Party: Sponsor
Other Study IDs: TD08-200
Record Dates: First submitted 2016-09-01; First posted 2016-09-12 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Solid Neoplasms
Keywords: neoplasms; hyperthermia
MeSH Terms: conditions — Neoplasms; Hyperthermia | interventions — Diathermy; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hyperthermia: treatment with the Celsius42 Hyperthermia System
  Interventions: Device: Hyperthermia

INTERVENTIONS:
Device: Hyperthermia — treatment with the Celsius42 Hyperthermia System additional to radiotherapy and/or chemotherapy
  Other Names: treatment with the Celsius42 Hyperthermia System

SUMMARY:
Based on the basic data of all patients foreseen for a local hyperthermia in the participating centers the failure rate (of the Celsius TCS Hyperthermia System) and the complication rate (injury to the patients) will be recorded.

DETAILED DESCRIPTION:
During this PMCF Trial from each participating center the internal data of all Celsius TCS Hyperthermia devices are collected. The participating centers are obligated to report any device-related failure and Adverse Event (injury to the patient). The center reports together with the device-internal data allows to calculate the failure and the complication rates. It will be analyzed regarding the kind of tumor and the concomitant treatment (radiotherapy and/or chemotherapy). The outcome groups (with/without failure or complication) will be analyzed regarding demographic and treatment parameters.

ELIGIBILITY:
Inclusion Criteria:

* treatment performed with the Celsius TCS Hyperthermia System

Exclusion Criteria:

* not applicable -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all treatments performed with the Celsius TCS Hyperthermia System at the participating centers throughout the study period. (Normally these are neoplasm patients treated additionally with radiation and/or chemotherapy.)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
failures of the device as well as failure of persons using the device during treatment | one month after treatment
  Based on the risk analysis the failures occurring during treatment will be classified and their frequency will be evaluated. This will be done using the investigators' judgment regarding severity of the failures (as minor, moderate, severe).
any injury, harm or medically relevant discomfort occurring for the patients or the staff | one month after treatment
  Based on the risk analysis the injuries occurring during treatment will be classified and their frequency will be evaluated. This will be done using the investigators' judgment regarding severity of the failures (as minor, moderate, severe).

CONTACTS AND LOCATIONS:
Overall Officials: Hüseyin Şahinbaş, MD, Principal Investigator — Praxis-Klinik Hyperthermie

IPD SHARING:
Plan to Share IPD: No